CLINICAL TRIAL: NCT04460885
Title: A 78-week Trial Comparing the Effect and Safety of Once Weekly Insulin Icodec and Once Daily Insulin Glargine 100 Units/mL, Both in Combination With Non-insulin Anti-diabetic Treatment, in Insulin naïve Subjects With Type 2 Diabetes
Brief Title: A Research Study to Compare Two Types of Insulin, a New Insulin, Insulin Icodec and an Available Insulin, Insulin Glargine, in People With Type 2 Diabetes Who Have Not Used Insulin Before
Acronym: ONWARDS 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4477; U1111-1247-3878 (Other: World Health Organization (WHO)); 2020-000442-34 (EudraCT Number)
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec (Experimental): Insulin icodec + non-insulin anti-diabetic drugs. The pre-trial non-insulin anti-diabetic background medication should be maintained at the stable, pre-trial dose and at the same frequency during the entire treatment period
  Interventions: Drug: Insulin icodec
- Insulin glargine (Active Comparator): Insulin glargine + non-insulin anti-diabetic drugs. The pre-trial non-insulin anti-diabetic background medication should be maintained at the stable, pre-trial dose and at the same frequency during the entire treatment period
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneous (s.c.) injections of insulin icodec once weekly for 78 weeks.
  Arms: Insulin icodec
Drug: Insulin glargine — Participants will receive subcutaneous (s.c.) injections of insulin glargine once daily for 78 weeks
  Arms: Insulin glargine

SUMMARY:
This study compares insulin icodec (a new insulin taken once a week) to insulin glargine (an insulin taken once daily which is already available on the market) in people with type 2 diabetes.

The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin glargine taken daily. Participants will either get insulin icodec that participants will have to inject once a week on the same day of the week or insulin glargine that participants will have to inject once a day at the same time every day. Which treatment participants get is decided by chance.

The insulin is injected with a needle in a skin fold in the thigh, upper arm or stomach. The study will last for about 1 ½ years. Participants will have 37 clinic visits and 26 phone calls with the study doctor. At 11 clinic visits participant will have blood samples taken. At 8 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Participants will be asked to wear a sensor that measures the blood sugar all the time in 5 periods of about one month during the study (about 5 months in total). Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus (T2D) 180 days or more prior to the day of screening.
* HbA1c from 7.0-11.0% (53.0-96.7 mmol/mol) both inclusive at screening confirmed by central laboratory analysis.
* Insulin naïve. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes.
* Stable daily dose(s) 90 days or more prior to the day of screening of any of the following anti-diabetic drug(s) or combination regimen(s): a. Any metformin formulations at least or greater than 1500 mg or maximum tolerated or effective dose. b. Any metformin combination formulations equal to or above 1500 mg or maximum tolerated or effective dose. c. Any of the following oral anti-diabetic drug classes including combinations ((equal to or above half of the maximum approved dose according to local label or maximum tolerated or effective dose): Sulfonylureas, Meglitinides (glinides), dipeptidyl peptidase-4 (DPP-4) inhibitors, Sodium-glucose co-transporter-2 (SGLT2) inhibitors, Thiazolidinediones, Alpha-glucosidase inhibitors, Oral combination products (for the allowed individual oral anti-diabetic drugs), Oral or injectable glucagon-like peptide 1 (GLP-1) receptor agonists
* Body mass index (BMI) equal to or below 40.0 kg/m^2.

Exclusion Criteria:

* Any episodes (as declared by the subject or in the medical records) of diabetic ketoacidosis within 90 days prior to the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (198):
- United States (97):
  - Uni of Alabama at Birmingham, Birmingham, Alabama
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Advanced Clinical Research/Rancho Paseo Medical Group, Banning, California
  - American Clinical Trials, Buena Park, California
  - San Fernando Valley Hlth Inst, LLC, Canoga Park, California
  - Med Center Medical Clinic, Carmichael, California
  - Headlands Research California, LLC, Escondido, California
  - Valley Research, Fresno, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - Clinical Trials Research_Sacramento, Lincoln, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Providence Clinical Research, North Hollywood, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - NorCal Endocrinology and Internal Medicine_Roseville, Roseville, California
  - Diabetes Research Center, Tustin, California
  - Coastal Metabolic Research Center, Ventura, California
  - Denver Endocrinology Diabetes and Thyroid Center, Englewood, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Revival Research, Doral, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Clinical Research of Cent FL, Winter Haven, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - RNA America Health Sciences, Sugar Hill, Georgia
  - East West Medical Research Institute_Honolulu, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Central Illinois Diabetes and Clinical Research, Springfield, Illinois
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - St Elizabeth Physicians Heart, Covington, Kentucky
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Endo And Metab Cons, Rockville, Maryland
  - Arcturus Healthcare, PLC., Troy, Michigan
  - Diabetes & Endo Specialists Inc, Chesterfield, Missouri
  - Methodist Phys. Clinic, Omaha, Nebraska
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern NH Diabetes and Endo_Nashua, Nashua, New Hampshire
  - Albuquerque Clin Trials, Inc., Albuquerque, New Mexico
  - N.Y. Total Medical Care PC, Brooklyn, New York
  - Northwell Health Div of Endo, Great Neck, New York
  - NYU Grossman School of Med, New York, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Medication Management, LLC, Raleigh, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - Clinical Research Source Inc, Perrysburg, Ohio
  - Intend Research, Norman, Oklahoma
  - Oregon Health & Science University_Portland, Portland, Oregon
  - Heritage Valley Medical Group Inc, Beaver, Pennsylvania
  - Indiana-Armstrong Endocrinology Associates, Indiana, Pennsylvania
  - The Diabetes Center, LLC, Murrells Inlet, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Texas Diab & Endo, P.A., Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - JCCT- Juno NW Houston, Houston, Texas
  - Fmc Science, Llc, Lampasas, Texas
  - Texas Diab & Endo, P.A., Round Rock, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Elite Medical Care, Sugar Land, Texas
  - Wade Family Medicine, Bountiful, Utah
  - Advanced Research Institute, Ogden, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Danville Internal Medicine Inc, Danville, Virginia
  - TPMG Clinical Research, Newport News, Virginia
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Croatia (4):
  - Poliklinika SLAVONIJA OSIJEK, Osijek, County of Osijek-Baranja
  - Opca bolnica Karlovac, Karlovac
  - KBC Rijeka, Endokrinologija, Rijeka
  - Opca bolnica Varazdin_Endocrinology, Varaždin
- India (12):
  - PGIMS Rohtak, Rohtak, Haryana
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - chelleram Diabetes Institute, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Gandhi Hospital & Medical college, Hyderabad, Telangana
  - Osmania General Hospital, Hyderabad, Telangana
  - Ramdev Rao Hospital, Hyderabad, Telangana
  - SSKM, Kolkata, West Bengal
- Israel (6):
  - Soroka MC - Outpatient Diabetes Clinic, Beersheba
  - Wolfson MC - Diabetes Clinic, Holon
  - Hadassah Ein Karam MC - Diabetes Unit, Jerusalem
  - Diabetes Clinic Meir MC, Kfar Saba
  - Rabin MC Beilinson - Department of Cardiothoracic Surgery, Petah Tikva
  - Kaplan MC - Metabolic Unit, Rehovot
- Italy (5):
  - Policlinico Umberto I Seconda Clinica Medica, Roma, RM
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - Ospedale Maggiore Policlinico UO Endocrinologia Diabetolgia, Milan
  - Policlinico Universitario Paolo Giaccone, Palermo
- Japan (15):
  - Hayashi Diabetes Clinic, Chigasaki-shi, Kanagawa, Kanagawa, Japan
  - Hayashi Diabetes Clinic_Internal Medicine and Diabetes Medicine, Chigasaki-shi, Kanagawa, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - The University of Tokyo Hospital, Diabetes and Metabolic, Bunkyo-ku, Tokyo
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Sugimoto Clinic,Internal Medicine, Kitakyusyu-shi, Fukuoka
  - Toranomon Hospital, Endocrinology and Metabolism, Minato-ku, Tokyo
  - Shinden Higashi Clinic_Miyagi, Miyagi
  - Takatsuki Red Cross Hospital_Diabetes and Endocrine Div., Osaka
  - Shimizu Clinic Fusa, Saitama
  - Wakakusa Clinic, Shimotsuke-shi, Tochigi
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Noritake Clinic, Ushiku-shi, Ibaraki
- Mexico (4):
  - InstitutoJalisciense de Investigación en Diabetes y Obesidad, Guadalajara, Jalisco
  - Clínica Omega Diabetes, S.C., Mexico City, México, D.F.
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
  - Investigación Médica Sonora S.C., Hermosillo, Sonora
- Poland (8):
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin, Lublin Voivodeship
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - NBR Polska Tomasz Klodawski, Warsaw, Masovian Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne "Diabetika", Radom
  - Centrum Zdrowia Tuchow Sp z o.o., Wierzchosławice
  - Prywatny Gabinet Janusz Gumprecht, Zabrze
- Puerto Rico (3):
  - Advanced Clinical Research LLC, Bayamón
  - Manati Ctr For Clin Research, Manatí
  - Consultorio Medico, San Juan
- Russia (14):
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Setchenov First Moscow State Medical University, Moscow
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - Scientifc Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Medinet LLC, Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Regional clinical cardiology dispensary, Saratov
  - Siberian State Medical University, Tomsk
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Slovakia (8):
  - Peter Farkas MD, s.r.o., Šahy, Slovak Republic
  - Amb. diabetologie a poruch latkovej premeny a vyzivy, Bratislava
  - Diacrin s. r. o., Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
  - MediVet s.r.o., Malacky
  - SIN AZUCAR s.r.o., Malacky
  - Diabetologicka ambulancia SchronerMED, s.r.o., Moldava nad Bodvou
  - ARETEUS s.r.o., Trebišov
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - ABS La Roca del Vallés_Endocrinología, La Roca Del Vallés
  - Hospital Universitario de la Princesa, Madrid
  - Centro de Especialidades José Marva, Madrid
  - Hospital Quirón, Pozuelo de Alarcón
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
- United Kingdom (16):
  - Bollington Medical Centre, Bollington, Cheshire
  - Layton Medical Centre, Blackpool
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Countess of Chester Hospital, Chester
  - The Adam Practice, Dorset
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Wycombe General Hospital, High Wycombe
  - Burbage Surgery, Hinckley
  - Queen Alexandra Hospital_Portsmouth, Portsmouth
  - The Staploe Medical Centre, Soham
  - Joint Clinical Research Facility - Swansea, Swansea
  - Royal Cornwall Hospital (Treliske), Truro
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Derived] Mohan V, Kesavadev J, Murthy LS, Anil G, Chandrappa M, Kar S, Mishra S. Efficacy and Safety of Once-Weekly Insulin Icodec in Indian Participants with Diabetes: Results from ONWARDS 1, 4, and 6 Studies. Diabetes Ther. 2025 Nov;16(11):2193-2212. doi: 10.1007/s13300-025-01799-4. Epub 2025 Oct 6. PMID 41051694
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Riddell MC, Heller S, Carstensen L, Rocha TMP, Kehlet Watt S, Woo VC. The effect of once-weekly insulin icodec vs once-daily basal insulin on physical activity-attributed hypoglycaemia in type 2 diabetes: a post hoc analysis of ONWARDS 1-5. Diabetologia. 2025 Jul;68(7):1416-1422. doi: 10.1007/s00125-025-06414-6. Epub 2025 Apr 5. PMID 40186685
- [Derived] Bergenstal RM, Asbjornsdottir B, Watt SK, Lingvay I, Mader JK, Nishida T, Rosenstock J. Continuous glucose monitoring-based metrics and the duration of hypoglycaemia events with once-weekly insulin icodec versus once-daily insulin glargine U100 in insulin-naive type 2 diabetes: an exploratory analysis of ONWARDS 1. Lancet Diabetes Endocrinol. 2024 Nov;12(11):799-810. doi: 10.1016/S2213-8587(24)00220-1. Epub 2024 Oct 4. PMID 39374601
- [Derived] Polonsky W, Benamar M, Carstensen L, Davies M, Meller Donatsky A, Franek E, Kellerer M, Philis-Tsimikas A, Goldenberg R. Improved treatment satisfaction with once-weekly insulin icodec compared with once-daily basal insulin in individuals with type 2 diabetes: An analysis of patient-reported outcomes and participant interviews from ONWARDS 2 and 5 and a physician survey from ONWARDS 1. Diabetes Res Clin Pract. 2024 Nov;217:111885. doi: 10.1016/j.diabres.2024.111885. Epub 2024 Oct 4. PMID 39368488
- [Derived] Watada H, Asbjornsdottir B, Nishida T, Nishimura R, Yamamoto Y, Yamauchi T, Kadowaki T. Efficacy and safety of once-weekly insulin icodec versus once-daily basal insulin in Japanese individuals with type 2 diabetes: A subgroup analysis of the ONWARDS 1, 2 and 4 trials. Diabetes Obes Metab. 2024 Dec;26(12):5882-5895. doi: 10.1111/dom.15960. Epub 2024 Sep 30. PMID 39344833
- [Derived] Rosenstock J, Bain SC, Gowda A, Jodar E, Liang B, Lingvay I, Nishida T, Trevisan R, Mosenzon O; ONWARDS 1 Trial Investigators. Weekly Icodec versus Daily Glargine U100 in Type 2 Diabetes without Previous Insulin. N Engl J Med. 2023 Jul 27;389(4):297-308. doi: 10.1056/NEJMoa2303208. Epub 2023 Jun 24. PMID 37356066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 137 sites in 12 countries while 141 sites screened participants. The total number of sites per country that screened and randomised participants are as follows (number of sites that screened participants/number of sites that randomised participants): Croatia (4/4), India (9/9), Israel (5/5), Italy (5/5), Japan (14/14), Mexico (3/3), Poland (8/8), Russia (14/14), Slovakia (7/7), Spain (5/5), United Kingdom (11/11), United States (56/52)
Groups:
- Insulin Icodec: Participants received once-weekly subcutaneous injection of insulin icodec at a starting dose of 70 U for 78 weeks using PDS 290 pre-filled injector in combination with non-insulin anti-diabetic drugs. The dose adjustment was based on the three pre-breakfast self-monitored plasma glucose (SMPG) values measured on two days prior to titration and on the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per liter (mmol/L): dose reduced by 20 units (U); 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 20 units.
- Insulin Glargine: Participants received once daily subcutaneous injection of insulin glargine at a starting dose of 10 U for 78 weeks using SoloSTAR pre-filled pen injector in combination with non-insulin anti-diabetic drugs. The dose adjustment was based on the three pre-breakfast self-monitored plasma glucose (SMPG) values measured on two days prior to titration and on the day of the contact. If atleast one pre-breakfast SMPG value was: < 4.4 mmol/L: the dose was reduced by 3 U; 4.4-7.2: no dose adjustment required and >7.2 mmol/L: dose was increased by 3 U.
Period: Overall Study
Arm/Group | Insulin Icodec | Insulin Glargine
Started | 492 | 492
Full Analysis Set | 492 | 492
Safety Analysis Set | 492 | 492
Completed | 474 | 475
Not Completed | 18 | 17
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Site closure | 1 | 0
Not completed — Death | 5 | 4
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec | Insulin Glargine | Total
Number analyzed (Participants) | 492 | 492 | 984
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.06 (10.05) | 58.85 (9.85) | 58.96 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 229 | 426
  Male | 295 | 263 | 558
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 53 | 106
  Not Hispanic or Latino | 439 | 439 | 878
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 129 | 145 | 274
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 10 | 17 | 27
  White | 333 | 317 | 650
  Other | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to week 52 is presented. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 52
Population: Full analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Percentage of HbA1c | -1.55 (0.06) | -1.35 (0.05)
Statistical Analysis 1: Comparison: Insulin Icodec vs Insulin Glargine; Test type: Non-Inferiority — The response and change from baseline in response after 52 weeks are analysed using an analysis of covariance (ANCOVA) model with treatment and region as fixed factors, and baseline response as covariate; p < 0.0001, ANCOVA; Treatment difference = -0.19, 95% CI 2-sided [-0.36 to -0.03]

2. Secondary Outcome: Percentage of Time in Target Range 3.9-10.0 mmol/L (70-180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time in target range 3.9-10.0 mmol/L (70-180 mg/dL) using CGM system from week 48 to week 52 is presented. Time in target range is defined as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive, divided by the total number of recorded measurements. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: From week 48 to week 52
Population: Full analysis set included all randomized participants. Overall number of participants analysed = Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 439 | 440
Percentage of time | 71.94 (18.23) | 66.90 (18.19)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline (week 0) to week 52 is presented. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 480 | 474
millimoles per liter (mmol/L) | -3.35 (0.09) | -3.33 (0.09)

4. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3) Until Week 52
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemic episode is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on main-on-treatment period. Main-on-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the end-date of the on-treatment period or week 52. On-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From baseline (week 0) to week 52
Population: Safety analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 1 | 3

5. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than [<] 3.0 mmol/L [54 mg/dL] Confirmed by Blood Glucose [BG] Meter) Until Week 52
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL) confirmed by BG meter) is presented. Clinically significant hypoglycaemia is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. The outcome data was evaluated based on main-on-treatment period. Main-on-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the end-date of the on-treatment period or week 52. On-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From baseline (week 0) to week 52
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 143 | 75

6. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3) Until Week 52
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) is presented. Clinically significant hypoglycaemia is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemic episode is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on main-on-treatment period. Main-on-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the end-date of the on-treatment period or week 52. On-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From baseline (week 0) to week 52
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 144 | 78

7. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3) Until Week 83
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemic episode is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on on-treatment period. The on-treatment period started at the date of first dose of trial product as recorded on the eCRF, and ended at the first date of any of the following: The end of trial visit (V63), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a subject was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 83
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 1 | 7

8. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL) Confirmed by BG Meter) Until Week 83
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL) confirmed by BG meter) is presented. Clinically significant hypoglycaemia is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. The outcome data was evaluated based on on-treatment period. The on-treatment period started at the date of first dose of trial product as recorded on the eCRF, and ended at the first date of any of the following: The end of trial visit (V63), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a subject was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 83
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 226 | 114

9. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3) Until Week 83
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) is presented. Clinically significant hypoglycaemia is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemic episode is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on on-treatment period. On-treatment period started at the date of first dose of trial product as recorded on the eCRF and ended at the first date of any of the following: The end of trial visit (V63), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. On-treatment period was the period in which a participant was exposed to trial product.
Time Frame: From baseline (week 0) to week 83
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Episodes | 227 | 121

10. Secondary Outcome: Mean Weekly Insulin Dose
Description: Mean weekly insulin dose from week 50 to week 52 is presented. The outcome data was evaluated based on main on treatment period. Main-on-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the end-date of the on-treatment period or week 52. On-treatment period started with onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From week 50 to week 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
Units of insulin | 214.23 [202.18 to 227.0] | 222.39 [209.93 to 235.59]

11. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 52 is presented. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 52
Population: Full analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 492 | 492
kilograms (kg) | 2.29 (0.21) | 1.83 (0.21)

12. Secondary Outcome: Percentage of Time Spent < 3.0 mmol/L (54 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent < 3.0 mmol/L (54 mg/dL) from week 48 to week 52 is presented. Time spent below threshold is defined as 100 times the number of recorded measurements below the threshold, divided by the total number of recorded measurements. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: From week 48 to week 52
Population: Full analysis set included all randomized participants. Overall number of participants analyzed=Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 439 | 440
Percentage of time | 0.27 (0.57) | 0.21 (0.63)

13. Secondary Outcome: Percentage of Time Spent > 10 mmol/L (180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent > 10 mmol/L (180 mg/dL) is presented. Time spent above threshold is defined as 100 times the number of recorded measurements above the threshold, divided by the total number of recorded measurements. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomization and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit), death for participants who died before any of the above.
Time Frame: From week 48 to week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 439 | 440
Percentage of time | 26.86 (18.74) | 32.27 (18.66)

ADVERSE EVENTS:
Time Frame: From week 0 to week 83
Description: Treatment emergent adverse events (TEAEs) are reported: event that had onset date during on-treatment period: started 1st dose date of trial product as recorded on eCRF, and ended at 1st date of any of following: end of trial V63, last date on trial product+5 weeks for once daily insulin and+6 weeks for once weekly insulin, end-date for in-trial observation period. Safety analysis set: all participants randomly assigned to trial treatment who took at least 1 dose of trial product.
Arm/Group | Insulin Icodec | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 5/492 | 4/492
Serious Adverse Events (participants affected / at risk) | 64/492 | 71/492
Other Adverse Events (participants affected / at risk) | 221/492 | 216/492
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=492) | Insulin Glargine (N=492)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 5 (5)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 4 (4) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (2) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Deafness traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrolyte depletion (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Immunisation reaction (Immune system disorders) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (2) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=492) | Insulin Glargine (N=492)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (36) | 22 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (42) | 32 (34)
COVID-19 (Infections and infestations) | 87 (91) | 101 (108)
Diabetic retinopathy (Eye disorders) | 36 (41) | 32 (38)
Diarrhoea (Gastrointestinal disorders) | 39 (54) | 26 (29)
Nasopharyngitis (Infections and infestations) | 38 (50) | 47 (56)
Pyrexia (General disorders) | 27 (30) | 23 (27)
Upper respiratory tract infection (Infections and infestations) | 28 (40) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT04460885/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT04460885/SAP_001.pdf